CLINICAL TRIAL: NCT00155116
Title: SERPIN D1 and Its Role in Lung Cancer Invasion and Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701095
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2004-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
To evaluate the correlation between SERPIN D1 expression in clinical specimen (including surgical specimen and blood sample) and lung cancer metastasis.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in Taiwan and world wild. Although there were progresses in the diagnosis and treatment of lung cancer, the incidence and mortality rate of lung cancer increased in recent years. In many cases, lung cancer is not diagnosed and treated until cancer cells have already invaded surrounding tissues and metastasized throughout the body. Only 15% of lung cancer patients were operable at presentation and about half of them had long term survival. The remaining almost died of metastatic disease. Detecting lung cancers when they are at their earliest stages, and identify cancers with metastatic potential will have a higher probability of truly curing the disease. Molecules that are expressed uniquely or at high level by tumor cells in comparison to normal tissues and that may be secreted into accessible fluids such as blood, urine, or sputum may be useful as lung cancer biomarkers. By using tools in SAGE Genie of Cancer Genome Anatomy Project (CGAP), we identified a secreted protein, SERPIN D1, as an overexpressed gene in non-small cell lung cancer as compared with normal lung and any other normal tissue. In an established panel of human lung adenocarcinoma cell lines with different invasive activities (CL1-0 cells and its sublines CL1-1, and CL1-5, in ascending order of activity), we detected that the expression of SERPIN D1 was higher in CL1-5 than in CL1-0 and CL1-1. According to our preliminary results, we hypothesize that SERPIN D1 may play a role in lung cancer invasion and metastasis and may serve as a serum biomarker for prognosis stratification. For this study, we are going to evaluate the potential correlation between SERPIN D1 expression in clinical specimen (including surgical specimen and blood sample) and lung cancer metastasis.

ELIGIBILITY:
Inclusion Criteria:

* non-small cell lung cancer patient, pathological proved

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-10; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Yu Liao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan